CLINICAL TRIAL: NCT02480400
Title: The Effect of Patient and Investigator Expectation on the Efficacy of Escitalopram in the Treatment of Patients With Major Depressive Disorder.
Brief Title: The Effect of Patient and Investigator Expectation on the Efficacy of Escitalopram in the Treatment Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abarbanel Mental Health Center (Other Government)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Principal Investigator, Yoram Barak, Director of Psychogeriatrics, Abarbanel Mental Health Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Lu-Pl-001
Record Dates: First submitted 2015-06-22; First posted 2015-06-24 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Major Depressive Disorder
Keywords: MDD; Escitalopram; Placebo
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Escitalopram; Dexetimide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Supported Escitalopram (Experimental): Escitalopram, with assessment visits at baseline, and weeks 2, 4, 6 and 8
  Interventions: Drug: Escitalopram
- Escitalopram (Active Comparator): Escitalopram, with assessment visits at baseline, week 4 and week 8, and a safety visit at week 2
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Escitalopram — Patients diagnosed with MDD and will fulfill the inclusion and exclusion criteria will start with escitalopram 10mg, according to the Summary of Product Characteristics. At week 2, patients with a baseline MADRS between 22 and 29 continue on 10mg, and patients with a baseline MADRS > 30 receive a fixed dose 20mg until the end of treatment.
  Other Names: Cipralex, Lexapro
  Arms: Supported Escitalopram
Drug: Escitalopram — Patients diagnosed with MDD and will fulfill the inclusion and exclusion criteria will start with escitalopram 10mg, according to the Summary of Product Characteristics. At week 2, patients with a baseline MADRS between 22 and 29 continue on 10mg, and patients with a baseline MADRS > 30 receive a fixed dose 20mg until the end of treatment.
  Other Names: Cipralex, Lexapro
  Arms: Escitalopram

SUMMARY:
To evaluate the effect of visit number, patient expectation, and rater expectation of the efficacy of escitalopram treatment in fixed doses of 10 and 20mg, based on baseline severity in patients with MDD.

DETAILED DESCRIPTION:
This study is designed to determined if trial design, in the form of the frequency of patient contact (assessment visit numbers) has an effect on the efficacy outcome after 8-week treatment with escitalopram.

The placebo response is a major issue in clinical trials for psychiatric disorders-and especially in the management of depression. Possible contributing factors to this problem include diagnostic misclassification, issues concerning inclusion/exclusion criteria, outcome measures' lack of sensitivity to change, measurement errors, poor quality of data entry and verification, waxing and waning of the natural course of depression, regression toward the mean phenomenon, patient and clinician expectations about the trial, study design issues, non-specific therapeutic effects, and high attrition.

Over the past few decades, researchers have attempted to reduce the placebo effect in a variety of ways. Unfortunately, approaches with very little or no benefit have included restricting enrollment to selected populations, rater training, requirement of same rater, and placebo lead-in phases. Some benefits, although often marginal, have been derived from standardizing diagnostic procedures, managing clinicians' overestimation of change, simplification of study visits and assessments, minimizing nonspecific, therapeutic effects, extending trial duration, reducing number of sites, increasing the sensitivity of outcome measures, and reducing the number of treatment arms.

Thus far, there has been no attempt to develop new study designs aimed at reducing the placebo effect.

We are proposing a novel study design, suitable for doubleblind, trials in mood disorders. This design is aimed at characterizing and identifying both the overall placebo response rate and the sample size required for such

ELIGIBILITY:
Inclusion Criteria:

1. Outpatients, men and women between 18 and 65 years of age (both extremes included)
2. DSM IV-TR criteria for a current MDE lasting between 3 and 12 months
3. Baseline MADRS total score > 22

Exclusion Criteria:

1. WHO-5 total score > 13 or a score > 3 on any single item of the WHO-5 (not revealed to the investigator)
2. Other primary or co-primary psychiatric disorder which is more distressful for the patient than MDDD, as evaluated by investigator
3. Patients with any history of mania/bipolar I disorder
4. Patients using medications which are contraindicated with the use of escitalopram
5. Known contraindication for the use of citalopram or escitalopram
6. Patients that have not responded to 2 or more treatments with an adequate dose of an antidepressant for an adequate time
7. Patients receiving formal behaviour therapy, or systematic psychotherapy
8. Unable to understand or read Hebrew and give written informed consent
9. Prominent suicidal ideation > 5 on item 10 (suicidal thoughts) of the MADRS]
10. Alcohol or substance dependence in the past 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2010-06; Primary Completion 2012-06 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Sheehan Disability Scale | Change from baseline to study completion by week 8.
  The Sheehan Disability Scale (Sheehan 1983) is a composite of three self-rated items designed to measure the extent to which three major sectors in the patient's life are impaired by panic, anxiety, phobic, or depressive symptoms. This scale has been used widely in psychopharmacology randomized controlled trials, particularly for panic disorder. This anchored visual analog scale uses spatiovisual, numeric, and verbal descriptive anchors simultaneously to assess disability across three domains: work, social life, and family life.

SECONDARY OUTCOMES:
Montgomery Åsberg Depression Rating Scale | Change from baseline to study completion in week 8.
  This is a 10-item checklist. Widely used in drug-treatment trials, mainly because of its particular sensitivity to treatment effects. Since there is a comparative lack of emphasis on somatic symptoms, the scale is useful for the assessment of depression in people with physical illness.

CONTACTS AND LOCATIONS:
Overall Officials: Yehuda Baruch, MD, MHA, Study Chair — Abarbanel MHC, Israel.
Locations (1):
- Abarbanel MHC, Bat Yam, Israel

REFERENCES:
- [Background] Gomeni R, Lavergne A, Merlo-Pich E. Modelling placebo response in depression trials using a longitudinal model with informative dropout. Eur J Pharm Sci. 2009 Jan 31;36(1):4-10. doi: 10.1016/j.ejps.2008.10.025. Epub 2008 Nov 8. PMID 19041717